CLINICAL TRIAL: NCT03758599
Title: Exercise in Anxiety and Posttraumatic Stress Disorders - a Randomized Controlled Clinical Pilot Trial
Brief Title: Exercise in Anxiety and Posttraumatic Stress Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaet Innsbruck (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 256912
Record Dates: First submitted 2018-10-11; First posted 2018-11-29 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Anxiety
Keywords: Anxiety Disorder; Posttraumatic Stress Disorder; Sports intervention
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Stair Climbing; Nordic Walking

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial with three arms for the comparison of the efficacy of a climbing exercise program, an aerobic exercise program and a social contact control group on symptoms of AD/PTSD, worry symptoms, quality of life, physical activity, health-related resources and affective responses in patients with AD or PTSD.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Climbing Exercise Group (Experimental): At the beginning of each session, a standardized body-centered, mind-setting warmup of ten minutes will take place. The general warm-up will be followed by climbing specific warm-up, which will consist of bouldering (20-30 minutes). Afterwards the rope climbing session will start. Climbing sessions also contain several sport-specific skill-development training sessions to familiarize the participants with gear and rope management, to acquire footwork and route finding, and to locate good belay spots and resting positions while climbing. At the end of the climbing session a short cool-down of five minutes will be executed.
  Interventions: Procedure: Climbing
- Aerobic Exercise Group (Experimental): As the climbing exercise group, the aerobic exercise group will start with a ten minutes body-centered, mind-setting warm-up, followed by 60 minutes of Nordic walking and five minutes cool down. A physiotherapist or sport scientist will instruct and guide the group. Nordic walking will be performed at a moderate pace at varying paths.
  Interventions: Procedure: Nordic Walking
- Social Contact Control Group (Active Comparator): Patients allocated to the social contact control group will receive the same amount of social interaction as the exercise groups. A physiotherapist or sport scientist will be present while participants watch movies with relevant content to disease followed by interactive group discussions. This group is required to control for the impact of social contact/support on AD/PTSD and secondary outcomes.
  Interventions: Procedure: Social Contact

INTERVENTIONS:
Procedure: Climbing — All interventions are identical in their duration. To fulfill the WHO guidelines of health enhancing activity (minimum 150 minutes of moderate exercise per week), two 75 minutes exercise sessions per week will take place. After meeting the inclusion criteria and after allocation to one of the three groups, patients will receive their timetable with the exercise or group session dates.
  Arms: Climbing Exercise Group
Procedure: Nordic Walking — All interventions are identical in their duration. To fulfill the WHO guidelines of health enhancing activity (minimum 150 minutes of moderate exercise per week), two 75 minutes exercise sessions per week will take place. After meeting the inclusion criteria and after allocation to one of the three groups, patients will receive their timetable with the exercise or group session dates.
  Arms: Aerobic Exercise Group
Procedure: Social Contact — All interventions are identical in their duration. To fulfill the WHO guidelines of health enhancing activity (minimum 150 minutes of moderate exercise per week), two 75 minutes exercise sessions per week will take place. After meeting the inclusion criteria and after allocation to one of the three groups, patients will receive their timetable with the exercise or group session dates.
  Arms: Social Contact Control Group

SUMMARY:
Aim: Aerobic and resistance exercise showed anxiolytic effects in clinical populations. Climbing could further enhance self-efficacy. Aim of the study is to examine whether climbing exercise and aerobic exercise, compared to social contact control, reduces symptoms of disease in out-patients with anxiety disorder (AD) and post-traumatic stress disorder (PTSD). Further analyses are aiming to reveal differences between climbing - and aerobic exercise.

Design: Randomized controlled clinical trial Participants: Thirty out-patients diagnosed with International Classification of Disease-Version 10 (ICD-10) (F40, F41, F43.1) for AD or PTSD.

Intervention: Out-patients will be assigned randomly to a climbing exercise group (a), aerobic exercise group (Nordic walking) (b) or social contact control group (c).

Measurements: Primary outcome is symptom severity in AD or Post Traumatic Stress Disorders. Further secondary outcomes are evaluated by psychological questionnaires assessing depression, worry symptoms, quality of life, self-efficacy and affective responses. Metabolites of neurotransmitters, immune-activation markers and anthropometric data will be additionally provided as secondary physiological outcomes.

Duration: Intervention duration is four weeks with 2 x 75 min for every group (climbing exercise, aerobic exercise, social contact control). Measurement points are set at the beginning (t1), at the end of the intervention (t2) and 3 (t3) and 6 (t4) months follow-up.

DETAILED DESCRIPTION:
The proposed research project is designed as a randomized controlled clinical trial with three arms. The efficacy of a climbing exercise program, an aerobic exercise program and a social contact control group on primary and secondary study outcome will be investigated (see Figure 1). Patients will be first screened by the outpatient-unit of the Department of Psychosomatics at the Medical University of Innsbruck or remitted through the treating staff network community. When assessed as eligible for the study, a group of up to ten out-patients will be randomly selected and invited to an informative meeting. Patients receive study information and time tables for their group attendances. The intervention will start within the following week and will end four weeks after beginning. Follow-up assessments will take place three and six months after intervention.

In addition to the AD/PTSD symptom screening, secondary study outcomes will be assessed:

* at study inclusion (t1)
* at the end of the intervention (t2)
* three months after the intervention (t3)
* six months after the intervention (t4)

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of Anxiety Disorder or Post Traumatic Stress Disorder: F40, F41, F43.1;
* age range: 18-65
* written informed consent
* stable medication (if needed) for at least 3 weeks

Exclusion Criteria:

* acute psychosis or suicidal behaviour
* medical contraindication to physical activity (assessed by a clinician)
* cognitive deficits
* problems with German language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (t1) Symptoms of Anxiety at four weeks (t2), three months after intervention (t3) and six months after intervention (t4) | 1 hour before intervention, after 672 hours, after 2328 hours, after 4488 hours
  Beck Anxiety Inventory (BAI; Beck & Steer, 1990) The BAI ranges from 0 and 63 points with lower points indicating less symptoms of anxiety
Change from Baseline (t1) Symptoms of Posttraumatic Stress Disorder at four weeks (t2), three months after intervention (t3) and six months after intervention (t4) | 1 hour before intervention, after 672 hours, after 2328 hours, after 4488 hours
  Post Traumatic Stress Disorder Checklist Civil Version (PCL-5; Weathers et al., 2013) The PCL-5 ranges from 0 and 80 points with lower points indicating less symptoms of PTSD The PCL-5 ranges from 0 and 80 points with lower points indicating less symptoms of Posttraumatic Stress Disorder

SECONDARY OUTCOMES:
Change from Baseline (t1) Depression at four weeks (t2), three months after intervention (t3) and six months after intervention (t4) | 1 hour before intervention, after 672 hours, after 2328 hours, after 4488 hours
  Beck Depression Inventory (BDI-II; Beck et al., 1996) The BDI-II ranges from 0 and 63 points with lower points indicating less symptoms of depression.
Change from Baseline (t1) Worry Symptoms at four weeks (t2), three months after intervention (t3) and six months after intervention (t4) | 1 hour before intervention, after 672 hours, after 2328 hours, after 4488 hours
  Penn-State Worry Questionnaire (PSWQ; Meyer et al., 1990) The PSWQ ranges from 16 and 80 points with lower points indicating less worries.
Change from Baseline (t1) Quality of Life (WHO) at four weeks (t2), three months after intervention (t3) and six months after intervention (t4) | 1 hour before intervention, after 672 hours, after 2328 hours, after 4488 hours
  Quality of life (WHOQOL-BREF; WHOQOL Group, 1998) The WHOQOL-BREF ranges from 5 and 130 points with lower points indicating less quality of life.
Change from Baseline (t1) Self Efficacy at four weeks (t2), three months after intervention (t3) and six months after intervention (t4) | 1 hour before intervention, after 672 hours, after 2328 hours, after 4488 hours
  General Self-Efficacy Scale (GSE; Schwarzer & Jerusalem, 1995) The GSE ranges from 4 and 40 points with lower points indicating less resources in self efficacy.
Affective Responses_a | 1 minute before each intervention, after 38 minutes, after 75 minutes
  Feeling Scale (FS; Hardy & Rejeski, 1989) The FS ranges from +5 to -5 points with lower points indicating low affective valence.
Affective Responses_b | 1 minute before each intervention, after 38 minutes, after 75 minutes
  Felt Arousal Scale (FAS; Svebak & Murgatroyd, 1985) The FAS ranges from 1 to 6 points with lower points indicating low level of arousal.
Affective Responses_c | 1 minute before each intervention, after 75 minutes
  The Positive and Negative Affect Scale (PANAS; Watson, Clark, & Tellegen, 1988) The PANAS measures two subscales, positive affect (points ranging from 10 to 50) and negative affect (points ranging from 10 to 50) Lower points on positive subscale indicates low level of positive affect, low points on negative affect subscale indicates low level of negative affect.
Affective Responses_d | 38 minutes after beginning of intervention
  Rating of Perceived Exertion (RPE; Borg, 1998)
Change from Baseline (t1) Analyses of neurotransmitter metabolites at four weeks (t2), three months after intervention (t3) and six months after intervention (t4) | 1 hour before intervention, after 672 hours, after 2328 hours, after 4488 hours
  tryptophan-kynurenine and the phenylalanine-tyrosine pathways
Change from Baseline (t1) Analyses of immune-activation markers at four weeks (t2), three months after intervention (t3) and six months after intervention (t4) | 1 hour before intervention, after 672 hours, after 2328 hours, after 4488 hours
  neopterin and pro-inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Sperner-Unterweger, Prof. MD, Principal Investigator — University Hospital of Psychiatry II, Department of Psychiatry, Psychotherapy and Psychosomatics, Innsbruck Medical University
Locations (1):
- University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bichler CS, Niedermeier M, Hufner K, Galffy M, Sperner-Unterweger B, Kopp M. Affective Responses to Both Climbing and Nordic Walking Exercise Are Associated With Intermediate-Term Increases in Physical Activity in Patients With Anxiety and Posttraumatic Stress Disorder - A Randomized Longitudinal Controlled Clinical Pilot Trial. Front Psychiatry. 2022 Jun 9;13:856730. doi: 10.3389/fpsyt.2022.856730. eCollection 2022. PMID 35757205